CLINICAL TRIAL: NCT05637463
Title: Reasons for Emergency Department Utilization and Readmission in Postoperative 90 Days: A Retrospective Analysis Based on the Hospital Information Management System
Brief Title: Reasons for Emergency Department Utilization and Readmission in Postoperative 90 Days
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma CEBECİ, Principal Investigator, Akdeniz University
Other Study IDs: 06
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-10

CONDITIONS: Surgery; Nursing Caries
Keywords: Surgery,; emergency department,; readmission
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — no intervention was made

SUMMARY:
The objective of this study was conducted to examine the reasons for patients' utilization of the emergency department and the rates of readmission in the first 90 days after surgery.

DETAILED DESCRIPTION:
Background: Postoperative readmission rates of patients have been important indicators in the evaluation of quality service delivery and cost-effectiveness. This study was conducted to examine the reasons for patients' utilization of the emergency department and the rates of readmission in the first 90 days after surgery.

Material and methods: The research is based on actual patient data in the hospital information management system. In the study, the data of patients who had undergone surgery between January 1, 2018, and December 31, 2018, and presented to the emergency department in the first 90 days after surgery were retrospectively analyzed. Patient data about the date of surgery, type of surgery, department performing the surgery, patient age, gender, type of anesthesia, the length of postoperative hospital stay, date of discharge, date, and reason for presenting to the emergency department, and discharge status (admission, referral, discharge, or death, etc.) recorded on the hospital information management system were evaluated in accordance with "the 18 HIPAA" standards.

ELIGIBILITY:
Inclusion Criteria:

* Undergone surgery between January 1, 2018, and December 31, 2018,
* Presented to the emergency department

Exclusion Criteria:

• Patients who do not meet the inclusion criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population of the study consisted of 1705 patients who had undergone surgery between January 1, 2018 and December 31, 2018 and presented to the emergency department within the first 90 days after discharge.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Identify the causes of preventable post-operative emergency utilization | January 1, 2018, and December 31, 2018,
  the reasons for patients' utilization of the emergency department after surgery

SECONDARY OUTCOMES:
Contribute to the strategic planning for quality health service delivery by determining the complaints and repeated admission rates by unit. | January 1, 2018, and December 31, 2018,
  the reasons for applying complaints on the basis of clinics

CONTACTS AND LOCATIONS:
Overall Officials: Fatma CEBECİ, Study Director — Akdeniz University; Songül Bişkin Çetin, Principal Investigator — Akdeniz University; Volkan Doğru, Principal Investigator — Akdeniz University; Mustafa Coşkun, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No